CLINICAL TRIAL: NCT03648229
Title: African Glaucoma Laser Trial
Acronym: AGLT
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Funding unavailable
Sponsor: West Virginia University (Other)
Collaborators: University of Pittsburgh (Other); University of Michigan (Other)
Responsible Party: Principal Investigator, Anthony Realini, Professor of Ophthalmology, West Virginia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AGLT
Record Dates: First submitted 2018-08-14; First posted 2018-08-27 (Actual); Last update posted 2021-06-21 (Actual); Status verified 2021-06

CONDITIONS: Open-angle Glaucoma
Keywords: glaucoma; laser; Africa
MeSH Terms: conditions — Glaucoma, Open-Angle; Glaucoma

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, active-controlled parallel-group design
Who Masked: Outcomes Assessor
Masking Description: Study personnel assessing IOP will be masked to treatment assignment during the first 12-month period and to all prior IOP measurements at every visit. IOP will be obtained using the iCare tonometer which provides an objective, digital reading.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- SLT (Experimental): The study eye will undergo 360-degree selective laser trabeculoplasty (SLT), followed, if needed, by repeat 360-degree SLT.
  Interventions: Procedure: Selective laser trabeculoplasty (SLT)
- MED (Active Comparator): The study eye will receive latanoprost ophthalmic solution 0.005% once daily, followed, if needed, by adjunctive timolol ophthalmic solution 0.5% twice daily. Medications will be provided at no cost to the subject.
  Interventions: Drug: Latanoprost ophthalmic solution; Drug: Timolol ophthalmic solution
- RX (Active Comparator): The study eye will receive latanoprost ophthalmic solution 0.005% once daily, followed, if needed, by adjunctive timolol ophthalmic solution 0.5% twice daily. Medications will be provided by prescription to be obtained at the subject's expense. This represents usual care for glaucoma in Africa and other regions of the world.
  Interventions: Drug: Latanoprost ophthalmic solution; Drug: Timolol ophthalmic solution

INTERVENTIONS:
Procedure: Selective laser trabeculoplasty (SLT) — Delivery of laser energy to the trabecular meshwork of the eye with the goal of reducing intraocular pressure
  Arms: SLT
Drug: Latanoprost ophthalmic solution — Prostaglandin analogue topical ophthalmic medication for reduction of intraocular pressure
  Arms: MED; RX
Drug: Timolol ophthalmic solution — Timolol ophthalmic solution 0.5% for reduction of intraocular pressure
  Arms: MED; RX

SUMMARY:
The AGLT is a prospective, multicenter, randomized study in which adult black Africans with treatment-naive open-angle glaucoma are assigned to therapy with selective laser trabeculoplasty (SLT), medications provided at no cost (MED), or medications provided by prescription for subjects to obtain at their own expense as per usual care (RX). The overall goal of the AGLT is to determine the best treatment strategy for newly-diagnosed open-angle glaucoma in Africa.

DETAILED DESCRIPTION:
This study is designed to test the hypothesis that the efficacy of SLT is non-inferior to medical therapy and the effectiveness of SLT is superior to medical therapy for glaucoma. This is a prospective, multicenter, active-controlled, parallel-group randomized trial. One eye per subject is included in this study and is randomized 1:1:1 to one of three treatment arms:

1. SLT arm (provided at no cost)

   1. Step 1: Initial 360 degree SLT
   2. Step 2: Repeat 360 degree SLT
2. MED arm (provided at no cost)

   1. Step 1: Latanoprost 0.005% once daily
   2. Step 2: Adjunctive timolol 0.5% twice daily
3. RX arm (Usual Care- dispensed by prescription to be obtained at subjects' expense)

   1. Step 1: Prescription for latanoprost 0.005% once daily
   2. Step 2: Prescription for adjunctive timolol 0.5% twice daily

Screening and baseline data are collected over two initial study visits. Baseline intraocular pressure (IOP) is determined and target IOP is calculated as a 20% reduction from baseline IOP and IOP < 22 mmHg. Following the initiation of step one of assigned therapy, subjects in the SLT arm will attend a Week 1 safety visit. All subjects will be seen at Month 1 for the first efficacy evaluation, then again at Month 3 and then every 3 months thereafter through 36 months of follow-up. Eyes with IOP above target IOP at two consecutive visits during the first 12 months will be deemed to have failed current therapy and are advanced to step 2 of assigned therapy:

* In the SLT arm, if step 1 (initial SLT) does not achieve or maintain target IOP, step 2 (repeat SLT) should be performed. One repeat SLT (two total) are allowed in the first 12 months following initial SLT; thereafter, SLT can be repeated as often as every 6 months.
* In the MED and RX arms, if step 1 does not achieve target IOP, latanoprost therapy should be continued and timolol added.

In all arms, if subjects fail step 2 of assigned therapy before Month 12, the subject is discontinued from study therapy, treated as deemed appropriate by site investigators, and continues to attend scheduled study visits and undergo safety-related study assessments. At Month 12, subjects in the SLT arm who have failed step 2 of therapy (repeat SLT) by Month 12 exit the study (as failure of 2 SLT treatments within 12 months indicates the subject is a poor candidate for further SLT). At Month 12, subjects in the MED and RX arms who are still active in the study (either still a success with Step 1 or 2 of assigned therapy; or failed step 2 but continue to attend study visits for safety assessment) will cross over to the SLT arm, discontinue medications, and undergo initial SLT. These subjects will attend a safety visit 1 week later and the first efficacy visit 1 month later. One repeat SLT (two total) is allowed in the first 12 months following initial SLT for those crossing over from the MED and RX arms; thereafter, SLT can be repeated as often as every 6 months.

The primary outcome measure is intraocular pressure, which will be assessed by study personnel masked to treatment assignment during the first 12 months and to all prior IOP measurements at every visit.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Male or female black African aged 18 years or older
4. Diagnosed with

   1. early or moderate open-angle glaucoma in one or both eyes (cup-disc ratio (CDR) < 0.9 and (if available) no glaucoma-related visual field loss in the central 10° on automated perimetry; or,
   2. if diagnosed with advanced glaucoma (CDR > 0.9 or glaucoma-related visual field loss within the central 10° on automated perimetry), meet at least one of the following criteria:

   i. Surgery is not available in the region of the study site; or ii. The subject is deemed not to be a candidate for surgery in the investigator's judgment; or iii. Surgery was offered and refused with no knowledge of this study.
5. Treatment-naïve: no prior treatment for open-angle glaucoma (including medications, laser, or glaucoma surgery) in both eyes
6. Untreated intraocular pressure >18 mmHg and <32 mmHg in the study eye at both baseline visits
7. Best-corrected visual acuity no worse than 20/400 in the study eye measured using Snellen's chart
8. Open iridocorneal angle (Shaffer Grade 3 or 4) with no more than 3 clock hours of peripheral anterior synechiae in both eyes
9. No contraindications to any of the study interventions
10. For females of reproductive potential: use of highly effective contraception for at least 1 month prior to screening and agreement to use such a method during study participation.

Exclusion Criteria:

1. Any glaucoma diagnosis other than open-angle glaucoma
2. Advanced stage glaucoma, defined as CDR > 0.9 or visual field loss within the central 10° on automated perimetry attributable to glaucoma (in the investigator's judgment)

   * The rationale for excluding subjects with advanced glaucoma is that these subjects would typically undergo surgery rather than laser or medical treatment. However, subjects with advanced stage glaucoma can be enrolled if any of the following three conditions are met:
   * Surgery is not available in the region of the study site; or
   * The subject is deemed not to be a candidate for surgery in the investigator's judgment; or
   * Surgery was offered and refused with no knowledge of this study In these cases, the subject would not undergo surgery regardless of participation in the study, and therefore should not be prevented from participation on this basis alone.
3. Currently or previously under treatment for glaucoma using medications, laser therapy or surgical interventions
4. Any corneal pathology that would preclude accurate assessment of IOP by rebound tonometry
5. Any non-glaucoma intraocular surgical procedure within the past 6 months
6. Contraindications to any of the study interventions

   * For SLT: no known absolute contraindications
   * For latanoprost: known hypersensitivity to any product ingredients
   * For timolol: bronchial asthma or history of such; severe chronic obstructive pulmonary disease; sinus bradycardia (<55 beats per minute); second or third degree atrioventricular block; overt cardiac failure; cardiogenic shock; hypersensitivity to any product ingredients
7. Pregnancy or lactation
8. Inability to attend all scheduled study visits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-09-01 (Estimated); Primary Completion 2022-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
12-month survival using Step 1 of assigned therapy | Month 12
  The proportion of eyes in each treatment group that achieve and maintain target IOP (minimum 20% reduction from baseline and IOP < 22 mmHg) through Month 12 using only Step 1 of therapy

SECONDARY OUTCOMES:
12-month survival using Step 1 +/- Step 2 of assigned therapy | Month 12
  The proportion of eyes in each treatment group that achieve and maintain target IOP (minimum 20% reduction from baseline and IOP < 22 mmHg) through Month 12 using Step 1 +/- Step 2 of therapy
Nature and incidence of treatment-emergent adverse events | Month 12
  Nature and frequency of adverse events reported in each treatment arm
Clinical utility of repeat SLT | Month 36
  Mean IOP at each time point following repeat SLT compared to initial SLT; nature and incidence of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Anthony D Realini, MD, Study Chair — West Virginia University Eye Institute

IPD SHARING:
Plan to Share IPD: No
To be determined by NIH Data Sharing Policy